CLINICAL TRIAL: NCT04830488
Title: Pilot Testing of the Body Image After Head and Neck Cancer Treatment (BIHNC) Program
Brief Title: Body Image After Head and Neck Cancer Treatment
Acronym: BIHNC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bethany Rhoten (Other)
Responsible Party: Sponsor-Investigator, Bethany Rhoten, Principal Investigator, Vanderbilt-Ingram Cancer Center
Organization: Vanderbilt-Ingram Cancer Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: VICC HN 2123
Record Dates: First submitted 2021-03-29; First posted 2021-04-05 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Head and Neck Cancer
Keywords: body image
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Body Image after Head and Neck Cancer Treatment (Experimental)
  Interventions: Behavioral: e-learning didactic module; Behavioral: Personal reflection activities

INTERVENTIONS:
Behavioral: e-learning didactic module — Participants utilize e-learning
Behavioral: Personal reflection activities — Participants complete questionnaires

SUMMARY:
This is a pilot study of the Body Image after Head and Neck Cancer Treatment Program [BIHNC]. It is a six-week, psychoeducational, web-based program that includes e-learning didactic modules and personal reflection activities for participants to complete.

DETAILED DESCRIPTION:
Specific Aim 1: To assess the feasibility and acceptability of [BIHNC] in patients who have completed treatment for head and neck cancer and who have body image concerns.

H1a: Eighty percent of enrolled study participants who complete baseline self-report measures will complete the BIHNC Program.

H1b: Eighty percent of study participants completing the BIHNC Program will rate it acceptable on the intervention evaluation form.

Specific Aim 2: To assess the preliminary efficacy of BIHNC for reducing body image concerns in patients who have completed treatment for head and neck cancer and who have body image concerns.

H2: Body image scores will improve from pre- to post- intervention

ELIGIBILITY:
Inclusion Criteria:

* Completion of any form of head and neck cancer treatment between 3 and 24 months previously at study enrollment
* Answer in the affirmative to at least one of two questions concerning dissatisfaction with the way their body looks or function
* Have clinically significant body image concerns as defined by (BIS score > 10)

Exclusion Criteria:

* Undergoing head and neck cancer treatment at time of study enrollment
* Cognitive impairment that would preclude ability to provide informed consent
* Unable to read text on a computer screen
* Not able to read and understand English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2021-04-05 (Actual); Primary Completion 2024-03-04 (Actual); Study Completion 2024-03-04 (Actual)

PRIMARY OUTCOMES:
Percentage of participants who complete program | Approximately 6 weeks
Percentage of participants who will rate program as acceptable | Approximately 6 weeks

SECONDARY OUTCOMES:
Percentage of participants with improvement in body image indicators | Approximately 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bethany Rhoten, PhD, Principal Investigator — Vanderbilt Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2022-02-04): https://cdn.clinicaltrials.gov/large-docs/88/NCT04830488/ICF_000.pdf